CLINICAL TRIAL: NCT05633589
Title: A Phase I/Ⅱ a Clinical Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Efficacy of Sc610 Cell Injection in the Treatment of Advanced Urinary System Tumors
Brief Title: A Clinical Study to Evaluate Safety, Tolerance, Pharmacokinetics and Efficacy of Sc610 Injection for Treating Advanced Urinary System Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hai Huang, Director of Department of Urology Surgery, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sc610-015-2022
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Malignant Tumor of Urinary System (Disorder)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Sc610 cell injection (Experimental): This trial is designed single arm. All the subjects enrolled will receive the experimental intervention: Sc610 cell injection.
  Interventions: Biological: Sc610 cell injection

INTERVENTIONS:
Biological: Sc610 cell injection — Peripheral blood mononuclear cells (PBMCs) obtained via apheresis are used for cell product preparation. PD-1 positive T cells are isolated from PBMCs, are transduced with lentivirus loaded with "enhanced receptor" and "amplification factor", and cell quantity are amplified. The obtained Sc610 is used for one-time intravenous infusion.

SUMMARY:
This is an phase I/IIa, open-lable, single-arm, single-dose escalation and multiple-dose extention clinical study of cell therapy designed to observe and evaluate the tolerance, the pharmacokinetic characteristics, the safety and the efficacy of Sc610 cell injection in the treatment of advanced tumor of urinary system.

DETAILED DESCRIPTION:
This study consists of two phases: the first phase will be the dose exploration phase (Phase I), followed by the dose extension phase (Phase II).

In phase I, 3 subjects are enrolled for 1st treatment group, starting with single dose of Sc610 cell injection of 5.0x10^8. If there is no dose limiting toxicity (DLT) observed, 3 subjects are enrolled into treatment groups successively in sequential order of: 1) group 2: Single dose of Sc610 1.5x10^9; 2) group 3: Single dose of Sc610 5x10^9; and 3) gorup 4: Single dose of Sc610 1.5x10^10.

Starting from the completion of Sc610 reinfusion for first subject of the 1st dose group, the subject will be observed for no less than one week. If no serious toxic and adverse events occurrs, Sc610 reinfusion for the second and third subjects will be performed. If no DLT occurrs by the 14th days after completion of reinfusion for the 3rd subject, The study will proceed to the next treatment group. If DLT is observed in 1/3 of enrolled subjects, another 3 subjects will be enrolled. In any of the dose groups, if ≤1/6 subjects have DLT, subject enrollment for the next treatment group will start. If DLT occurs in ≥2/6 of subjects, the number of subjects in the previous dose group shall be reviewed. If there were only 3 subjects, 3 more subjects will be enrolled. If DLT occurs in ≤1/6 subjects, the dose will be defined as the maximum tolerable dose (MTD), and the dose escalation phase of the study will be completed. If DLT occurs in ≥2/6 subjects in the first dose group, a dose reduction exploration will be performed or the study will be terminated upon decision made by the Safety Committee.

In phase II, If no dose limiting toxicity event occurred upon the completion of treatment in each of the 4 groups. Researcher will decide to select 2-4 dose groups for dose extension study and will enroll 5-8 subjects for each group.

Certain subjects have the option to receive multiple rounds of Sc610 treatment: 1) Subjects with unconfirmed disease progression (non iCPD, i.e. iUPD, iSD, iPR) as assessed by the response to the cell treatment by medical imaging of last round of treatment can enter multiple rounds of treatment. Subjects with complete remission (iCR) will be allowed to receive one consolidation treatment；Subjects whose response to the cell treatment as assessed by medical imaging are disease progression (iCPD), and the investigator judge that the subjects would be unable to benefit from the treatment of this study, and need to receive a new treatment or change the treatment method, will fall off/withdraw from the trial. 2) Before entering the next round of treatment each time, the percentage of PD-1+T cells in total T cells need to be assayed first, and peripheral blood monocytes apheresis can be performed if the detection result is≥18% (PBMCs≥3 x10^9). The procedures of preparation, reinfusion, and follow-ups after reinfusion of Sc610 cell injection are the identical as before. 3) If toxic reaction related to Sc610 greater than grade 3 cells is observed in previous dose (round) of treatment, the dose of next round will be reduced; If adverse events above grade 3 still occur after dose reduction, the investigator will make a comprehensive judgment on whether to terminate the study of this subject. 4) Multiple round treatment is a treatment cycle every 12 weeks. After treatment, follow up until the disease progresses, or start a new anti-tumor treatment, or fall off, or withdraw from the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender;
2. Expected survival >3 months;
3. The physical condition score of the Eastern American Oncology Collaboration Group (ECOG) equal to 0 or 1;
4. Patients with pathologically confirmed, locally advanced, or recurrent metastatic advanced urinary system malignant tumors, failed in standard treatment, disease development after multi-line treatments, and cannot be surgically removed, including:

   1. Renal cell carcinoma: clear cell carcinoma, papillary renal cell carcinoma, chromophobe cell carcinoma, etc;
   2. Urothelial carcinoma: including renal pelvis, ureter, bladder, or urethra orginated;
   3. Prostate adenocarcinoma.
5. According to iRECIST standard, there exists at least one measurable tumor lesion as shown by CT or MRI. Measurable tumor lesions are defined as the longest diameter ≥10mm and scanning thickness ≤ 5.0mm. For lymph node lesions, the short diameter ≥ 15mm;
6. The proportion of peripheral blood PD-1+T cells in total T cells ≥ 18%; and voluntarily accept the apheresis of peripheral blood mononuclear cells for the preparation of Sc610 cell injection;
7. Sufficient bone marrow and organ functions:

   1. Hematology: neutrophils is equal to or higher than 1.5×10^9/L, platelets is equal to or higher than 75×10^9/L, hemoglobin is equal to or higher than 80g/L; total lymphocytes is equal to or higher than 60% of the lower limit of normal range;
   2. Hepatic function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are both eqal to or lower than 3 times the upper limit of normal range (ULN) (if intrahepatic bile duct cancer exists, equal to lower than 5 times of ULN); total bilirubin (TBIL) is equal to or lower than 1.5 times of ULN;
   3. Renal function: Creatinine (Cr) is equal to or lower than 1.5 times of ULN;
   4. Coagulation function: prothrombin time (PT) is equal to or shorter than 1.5 times of ULN or activated partial prothrombin time (APTT) is equal to or shorter than1.5 times of ULN;
8. Qualified patients with fertility (male and female) must agree to use reliable contraceptive methods (hormone or barrier method or abstinence, etc.) with their partners during the trial and at least 90 days after the last medication; The blood or urine pregnancy test within 7 days before the first administration of the study drug in women of childbearing age (From menarche to 1 year starting from menopause is considered fertile) must be negative;
9. Subjects need to be informed of this study before the trial, and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Intracranial metastasis or meningeal metastasis with clinical symptoms, or other evidence indicating that the intracranial metastasis or meningeal metastasis of the patient has not been controlled, and the vertebral body metastasis that is known or suspected to cause spinal cord compression, with which the investigator judge that the patient is not suitable for study enrollment;
2. Patients who have had or are currently suffering from other malignant tumors within 2 years before signing the contract, excluding cured patients with basal cell skin cancer, in situ cervical carcinoma, and in situ lung cancer;
3. Patients treated with PD-L1 monoclonal antibody (including but not limited to atezolizumab and duvalizumab) within 12 weeks before collection;
4. Those who have active infection within one week before single collection and need systematic anti infection treatment at present ;
5. People with interstitial lung disease ;
6. Patients who have received immunotherapy and have ≥ grade 3 IRAE;
7. Patients with active or ever suffered from autoimmune diseases with the possibility of recurrence (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except patients with clinically stable autoimmune thyroid diseases and well controlled type I diabetes ;
8. The adverse reaction of previous anti-tumor treatment has not recovered to CTCAE 5.0 grade evaluation ≤ 1 (except for the toxicity that the researcher judges is without risk for safety);
9. Have received anti-tumor treatment within 2 weeks before apheresis, including but not limit to systemic chemotherapy, radiotherapy, immunotherapy, etc; Nitrosourea or mitomycin C is defined within 6 weeks before apheresis;
10. Have received systemic glucocorticoid (prednisone ≥ 10mg/day or equivalent dose of the same type of drug) or other immunosuppressants within 2 weeks before apheresis; The following conditions are exempted: intermittent use of glucocorticoids in local, eye, joint cavity, nose, and inhalation; and short term use of glucocorticoid for preventive treatment (such as prevention of contrast agent allergy);
11. Have received other unlisted clinical research drugs or treatments within 4 weeks before apheresis;
12. Hepatitis B: HBsAg (+) or HbeAg (+); Or anti HBe (+)/anti HBc (+), and the hepatitis B DNA quantitation is higher than the lower detection limit of the research center; Hepatitis C: Anti HCV positive; Positive Treponema pallidum antibody; Positive HIV antibody test;
13. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limit to:

    1. Serious cardiac arrhythmia or conduction bockade, such as ventricular arrhythmia requiring clinical intervention, Ⅱ-Ⅲ degree atrioventricular blockade, etc;
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other cardiovascular and cerebrovascular events ≥Level 3 occurred within 6 months before the first study drug administration;
    3. New York Heart Association (NYHA) cardiac function classification ≥ Grade II or left ventricular ejection fraction (LVEF)≤50%, or with other structural heart disease that researchers judge as with high risk;
    4. Hypertension beyond clinical control.
14. The serous cavity effusion that cannot be controlled clinically is not suitable for the group according to the judgment of the investigator;
15. Known alcohol or drug dependence;
16. Mental disorders or poor compliance;
17. Pregnant or lactating women;
18. The investigator believes that the subject has a history of other serious systemic diseases or is not suitable to participate in this clinical study for other reasons.The adverse reaction of previous anti-tumor treatment has not recovered to CTCAE 5.0 grade evaluation ≤ 1 (except for the toxicity without safety risk judged by researchers such as hair loss);
19. Patients with active or had autoimmune diseases that may recur (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.); Except for patients with clinically stable autoimmune thyroid disease and well controlled type I diabetes;
20. Have a history of immunodeficiency, including HIV antibody test positive;
21. Hepatitis B (immunological test results do not exclude infectivity) and/or hepatitis B DNA titer is higher than the lower limit of the detection value of the research center; And/or hepatitis C (anti HCV antibody positive); And/or treponema pallidum antibody positive;
22. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    1. There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, ⅱ - ⅲ degree atrioventricular blockade, etc;
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events ≥ grade 3 occurred within 6 months before the cell reinfusion;
    3. New York Heart Association (NYHA) cardiac function rating ≥ class II or left ventricular ejection fraction (LVEF) <50%, or other structural heart disease with high risk as judged by the investigator;
    4. Clinically uncontrollable hypertension;
23. Serous cavity effusion beyond clinical control is not suitable for the enrollment according to the judgment of the investigator;
24. Known alcohol or drug dependence;
25. Mental disorders or poor compliance;
26. Pregnant or lactating women;
27. The investigator believes that the subject has a history of other serious systemic diseases or is not suitable to participate in this clinical study due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 weeks after single dose of cell reinfusion
  Including cases of complete response (CR) and of partial response (PR).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 12 weeks after the single dose of cell reinfusion
  The number of cases with remission and stable lesions after treatment accounted for the total number of evaluable cases.
Duration of Response (DOR) | 12 weeks after single dose of cell reinfusion
  Time from CR or PR to disease progression (PD), death, or last tumor evaluation.
Progression-Free Survival (PFS) | 12 weeks after single dose of cell reinfusion
  From the beginning of cell therapy to the time of the first disease progression or death due to any cause.
Overall survival (OS) | From single dose of cell reinfusion to death
  Time from cell reinfusion to death due to any cause
Adverse events (AEs) | 24 weeks after single dose of cell reinfusion
  According to National Cancer Institute Common Terminology Criteria for Adverse Events V5.0(CTCAE V5.0)
Detection of Lentivirus Copy Number | 12 weeks after single dose of cell reinfusion
  Dynamic changes of carrier gene copy number in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Hai Huang, Dr., Principal Investigator — Department of Urology Surgery, Sun Yat-sen Memorial Hospital of Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No